CLINICAL TRIAL: NCT01412658
Title: Safety Study of Milk Peptide Supplementation in Healthy Volunteers: a Randomized Placebo Controlled Clinical Trial
Brief Title: Clinical Safety of a Novel Milk Protein Peptide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ambryx Biotechnology (Industry)
Collaborators: Texas A&M University (Other); Baylor University (Other)
Responsible Party: Richard B Kreider, PhD, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AX_Safety_study
Record Dates: First submitted 2011-08-07; First posted 2011-08-09 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Drug Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Milk Peptides (Experimental)
  Interventions: Dietary Supplement: Hydrolyzed milk protein mixture
- Placebo (Placebo Comparator): Participants ingested 6ml - 21ml (based on participants' weight) of clear, sugar-less liquid placebo mixed with 1/2 cup milk twice daily (once immediately after breakfast and once immediately after dinner). The supplements were prepared in liquid form and packaged in generic bottles for double blind administration. The placebo was a glycerol-based placebo matched for color, texture, and taste to the active supplement.
  Interventions: Dietary Supplement: Glycerol placebo

INTERVENTIONS:
Dietary Supplement: Hydrolyzed milk protein mixture — Take twice a day, dosage 6 ml-21 ml based on weight, mix with 1/2 cup of milk.
  Other Names: AX-4
  Arms: Milk Peptides
Dietary Supplement: Glycerol placebo — Participants ingested 6ml-21ml of placebo mixed with 1/2 cup milk twice daily. The supplements were prepared in liquid form and packaged in generic bottles for double blind administration. The placebo was a starch-based placebo matched for color, texture, and taste to the active supplement.
  A food diary is maintained daily.
  Arms: Placebo

SUMMARY:
Background: A novel milk peptide has been shown in laboratory setting to have natural anti-cancer properties and extend lifespan and improve metabolism in animal models. The purpose of this study was 1.) to determine the safety dosage range and, 2.) to determine whether this novel milk peptide positively influence blood markers, metabolism and improve quality of life.

DETAILED DESCRIPTION:
The study was conducted as a randomized, double-blind, placebo-controlled clinical trial in a university research setting. Healthy volunteers were randomly assigned to ingest in a double-blind and randomized manner either a placebo or milk peptides. Outcome measures were assessed at 0, 3, and 6 weeks of supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with body mass index between 27-40.

Exclusion Criteria:

* have any metabolic disorders including known electrolyte abnormalities, heart disease, arrhythmias, diabetes, thyroid disease or hypogonadism; a history of hypertension, hepatorenal, musculoskeletal, autoimmune, or neurologic disease; if they are taking thyroid, hyperlipidemic, hypoglycemic, anti-hypertensive, or androgenic medications;
* have milk allergies

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2006-11; Primary Completion 2007-01 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Blood and Hormones | 6 weeks
  General whole blood and serum clinical chemistries (cholesterol, triglycerides, glucose, blood urea nitrogen, creatinine, uric acid, muscle and liver enzymes) and hormones (insulin, homeostasis model of insulin sensitivity, and leptin).

SECONDARY OUTCOMES:
Psychosocial | 6 weeks
  quality of life indices
Body Composition | 6 weeks
  All participants were tested for changes in energy intake and body composition

CONTACTS AND LOCATIONS:
Overall Officials: Rick Kreider, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Baylor University Center for Exercise, Nutrition, and Preventive Health Research, Waco, Texas, United States

REFERENCES:
- [Derived] Kreider RB, Iosia M, Cooke M, Hudson G, Rasmussen C, Chen H, Mollstedt O, Tsai MH. Bioactive properties and clinical safety of a novel milk protein peptide. Nutr J. 2011 Sep 26;10:99. doi: 10.1186/1475-2891-10-99. PMID 21943352
- See also: Exercise & Sport Nutrition Lab — http://exerciseandsportnutritionlab.com/